CLINICAL TRIAL: NCT00909350
Title: Micro-RNA (miR) Expression in Upper Gastrointestinal Mucosal Tissue: A Potential Target for Understanding and Preventing the Progression of Barrett's Esophagus
Brief Title: Micro-RNA (miR) Expression in Upper Gastrointestinal Mucosal Tissue
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kenneth R. DeVault, M.D., Professor and Chair, Department of Medicine, Mayo Clinic, Jacksonville Florida, Mayo Clinic
Other Study IDs: 06-005272
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Barrett's Esophagus; Esophageal Adenocarcinoma
Keywords: Barrett's esophagus; BE; esophageal adenocarcinoma; Micro-RNA; miR expression
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsy tissue from proximal and distal esophagus, stomach and duodenum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment: genetic research project; to meet inclusion criteria, participants must have normal upper GI tract upon upper endoscopy, for study biopsies to be taken

SUMMARY:
This is a laboratory-based, exploratory study using tissue obtained from our clinical practice. The purpose of this study is to confirm our ability to characterize miR expression in various tissues (proximal and distal esophagus, stomach and duodenum) obtained from the upper gastrointestinal tract in preparation for the study of MiR in patients with Barrett's esophagus and other inflammatory conditions of the upper gastrointestinal tract.

DETAILED DESCRIPTION:
The incidence of esophageal adenocarcinoma has increased dramatically over the past three decades. These adenocarcinomas usually arise from columnar lined epithelium of the esophagus known as Barrett's esophagus (BE). There is an established association between gastroesophageal reflux disease (GERD) and the development of BE and esophageal adenocarcinoma. In an attempt to diagnose esophageal adenocarcinoma at an earlier and more treatable stage, efforts have been directed at identifying patients with BE and enrolling them in surveillance protocols. Several authors have challenged this strategy since it has not yet been proven to save lives and is very expensive. A major unresolved problem is the fact that the clinical factors considered to be somewhat predictive of the presence or absence of BE are neither sufficiently sensitive nor specific. In addition, once BE is identified, predicting who may or may not progress to cancer is far from perfect. A molecular understanding of why certain patients develop BE and why certain of those progress to cancer is of obvious importance.

The molecular pathway from normal esophageal mucosa to Barrett's esophagus and on to adenocarcinoma is not well understood. Micro-RNA (miR) RNAs have recently emerged as important regulators of carcinogenesis and have not been studied in BE. We seek to confirm our ability to characterize miR expression in various tissues (esophagus, stomach and duodenum) obtained from the upper gastrointestinal tract in preparation for the study of MiR in patients with Barrett's esophagus and other inflammatory conditions of the upper gastrointestinal tract.

This study will involve collection of tissue via endoscopic biopsy in 10 patients with normal endoscopic appearance from the esophagus, stomach and duodenum. Ambion miR oligonucleotide arrays will be utilized to profile miRs that are specifically expressed in epithelial biopsies from the duodenum, stomach, and esophagus. Total RNA will be extracted from independent biopsy samples using the mirVana(R) micro RNA isolation kit from Ambion. The Ambion Flash PAGE(R) electrophoresis system will be used to resolve mature miRs from the larger pre-miR species. Mature miRs will be labeled and hybridized to Ambion mirVana miR(R)arrays, which will be scanned to identify miRs that are regulated under these circumstances. Signals from the microarrays will be processed using the R functions of Bioconductor for normalization and background correction and RMA for summarization. Statistical significance will be determined using Insightful S+ functions and assuming a least pooled error model. Potential targets will be confirmed by northern blotting. The routine histology sample will be reviewed simply to exclude other, unexpected microscopic pathology. Benign histologic findings such as minor inflammation, will not exclude the patient from inclusion. If there is a wide variation in miR expression, then the histology might be needed to help explain such variation.

ELIGIBILITY:
Inclusion Criteria:

* willingness to give consent
* normal gross appearance of the esophagus, stomach and duodenum

Exclusion Criteria:

* contraindication to mucosal biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects identified from individuals referred for upper endoscopy at Mayo Clinic in Jacksonville, Florida
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
miR expression between tissue from Barrett's esophagus and that from normal tissues | time it takes to have standard of care biopsies taken during one routine Upper Endoscopy

SECONDARY OUTCOMES:
expression of miR in Barrett's esophagus patients with cancer in comparison to those who do not progress to cancer | time it takes to have standard of care biopsies during one routine Upper Endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth R. DeVault,, M.D., Principal Investigator — Mayo Clinic, Jacksonville, Florida
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States